CLINICAL TRIAL: NCT01857141
Title: Comparative Study on the Effects of Epidural Dexmedetomidine on Heart Rate Variability During General Anesthesia in Patients Undergoing Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4-2011-0904
Record Dates: First submitted 2013-05-12; First posted 2013-05-20 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Gastric Cancer
Keywords: dexmedetomidine; heart rate variability; preemptive epidural; gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental)
  Interventions: Drug: preemptive dexmedetomidine epidural bolus injection(1.5 mcg/kg)
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: preemptive dexmedetomidine epidural bolus injection(1.5 mcg/kg) — Patients in the pre-emptive groups recived a dose of 1.5㎍/kg dexmedetomidine dissolved into normal saline 10cc before the induction of
  Arms: dexmedetomidine
Drug: normal saline — patients in the control groups received the equivalent volume of normal saline.
  Arms: normal saline

SUMMARY:
The use of epidural dexmedetomidine decreases the anaesthetic requirements and improved postoperative pain. Dexmedetomidine is a potent and highly selective a2-adrenoceptor agonist and has sympatholytic effect. Power spectral analysis of heart rate variability(HRV) is a useful tool to assess cardiac autonomic activity. We investigated whether preemptive epidural dexmedetomidine can develop hemodynamic change and it could be identify patients by HRV.

ELIGIBILITY:
Inclusion Criteria:

* Patients consented to spinal anesthesia were enrolled
* Patients aged 40~70 years olds undergoing gastrectomy
* No contraindication of epidural analgesia
* ASA class I and II
* Patients consented to epidural anesthesia were enrolled

Exclusion Criteria:

* Patients with hypovolemia, coagulation disorders, local infection at the site of operation, history of headache, heart diseases, and history of allergy, chronic alcohol use or abuse, anemia, congenital heart diseases, bundle block, congestive heart failure or arrythmias
* patients who had recently received sedative drugs or were under antidepressant treatment were not included in the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Heart rate variability analysis | 5min perioids after fluid resuscitation.
  Heart rate variability analysis was performed according to the Task Force recommendations.
  Frequency domain analysis was based on fast Fourier transformation. Power spectrum densities were calculated for low frequencies (LF: 0.04-0.15 Hz) and high frequencies (HF: 0.15-0.4 Hz) informalized units, defined as the LF or HF proportional part of the total power.
  Baseline and 30min after the injection of the study drug.

SECONDARY OUTCOMES:
Epidural injection | at 30 min after the epidural injection of the study drug
  And secondary data collection was done at 30 min after the epidural injection of the study drug.
  All of the HRV analysis was done before anaesthesia induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, Korea, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Bajwa SJ, Bajwa SK, Kaur J, Singh G, Arora V, Gupta S, Kulshrestha A, Singh A, Parmar S, Singh A, Goraya S. Dexmedetomidine and clonidine in epidural anaesthesia: A comparative evaluation. Indian J Anaesth. 2011 Mar;55(2):116-21. doi: 10.4103/0019-5049.79883. PMID 21712865
- [Background] Chatzimichali A, Zoumprouli A, Metaxari M, Apostolakis I, Daras T, Tzanakis N, Askitopoulou H. Heart rate variability may identify patients who will develop severe bradycardia during spinal anaesthesia. Acta Anaesthesiol Scand. 2011 Feb;55(2):234-41. doi: 10.1111/j.1399-6576.2010.02339.x. Epub 2010 Nov 8. PMID 21058941
- [Background] Hanss R, Bein B, Weseloh H, Bauer M, Cavus E, Steinfath M, Scholz J, Tonner PH. Heart rate variability predicts severe hypotension after spinal anesthesia. Anesthesiology. 2006 Mar;104(3):537-45. doi: 10.1097/00000542-200603000-00022. PMID 16508402
- [Background] Penttila J, Helminen A, Anttila M, Hinkka S, Scheinin H. Cardiovascular and parasympathetic effects of dexmedetomidine in healthy subjects. Can J Physiol Pharmacol. 2004 May;82(5):359-62. doi: 10.1139/y04-028. PMID 15213737
- [Background] Schnaider TB, Vieira AM, Brandao AC, Lobo MV. [Intraoperative analgesic effect of epidural ketamine, clonidine or dexmedetomidine for upper abdominal surgery.]. Rev Bras Anestesiol. 2005 Oct;55(5):525-31. doi: 10.1590/s0034-70942005000500007. Portuguese. PMID 19468643